CLINICAL TRIAL: NCT05191693
Title: Long-term Outcomes of Endoscopic Papillary Balloon Dilation for 8-12mm Bile Duct Stones: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Venizelio General Hospital (Other)
Responsible Party: Principal Investigator, Gregorios Paspatis, director of the gastroenterology department of Venizelio General Hospital, Venizelio General Hospital
Other Study IDs: Paspatis-balloon dilation
Record Dates: First submitted 2021-12-17; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Endoscopic Papillary Balloon Dilation; Bile Duct Stones; Endoscopic Sphincterotomy; Stone Recurrence
Keywords: endoscopic papillary balloon dilation; Stone recurrence
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with CBD stones up to 8-12mm: 72 patients (mean age: 67 years, 52.8% males) were included, of whom 22 (30.5%) had multiple CBD stones, 23 (31.9%) had a history of cholecystectomy, 13 (18.1%) had a periampullary diverticulum and 22 (30.5%) had a previous EST
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — endoscopic papillary balloon dilation (EPBD) with endoscopic sphincterotomy (EST
  Other Names: endoscopic papillary balloon

SUMMARY:
The investigators prospectively evaluated long-term outcomes of ELBPD+EST for CBD stones up to 8-12mm.

EPBD+EST in patients with CBD stones up to 8-12mm appears to be associated with a very low (<3%) rate of long-term stone recurrence. The efficacy of EPBD for 8-12mm stones warrants further exploration in randomized trials.

DETAILED DESCRIPTION:
Consecutive patients with CBD stones up to 8-12mm successfully treated by EPBD+EST from September 2018 to August 2020 were prospectively followed for at least 12 months. CBD stone recurrence was defined as recurrent stones confirmed by ERCP during the follow-up period. The maximum diameter of the balloon used was 15mm.

Overall, 72 patients (mean age: 67 years, 52.8% males) were included, of whom 22 (30.5%) had multiple CBD stones, 23 (31.9%) had a history of cholecystectomy, 13 (18.1%) had a periampullary diverticulum and 22 (30.5%) had a previous EST. The mean CBD diameter was 11.6±1mm, whereas a tapered duct was noted in 7 (9.7%). Post-procedural bleeding occurred in one case, treated successfully a with a fully covered metal stent. Mild cholangitis occurred in two cases. No cases with perforation or PEP were observed. During a mean follow-up of 22.4±6.2 months (range 13-36), CBD stones recurred in 2/72 (2.7%).

EPBD+EST in patients with CBD stones up to 8-12mm appears to be associated with a very low (<3%) rate of long-term stone recurrence. The efficacy of EPBD for 8-12mm stones warrants further exploration in randomized trials.

ELIGIBILITY:
Inclusion Criteria:patients with ELBPD+EST for CBD stones up to 8-12mm from September 2018 to August 2020 -

Exclusion Criteria: Patients with bile duct stones less than 8mm or more than 12mm.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with CBD stones up to 8-12mm successfully treated by EPBD+EST from September 2018 to August 2020 ,who were prospectively followed for at least 12 months
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Stone recurrence after endoscopic papillary balloon dilation (EPBD) with endoscopic sphincterotomy (EST) in prior ERCP. | 22.4±6.2 months
  Patients with CBD stones up to 8-12mm successfully treated by EPBD+EST from September 2018 to August 2020 were prospectively followed for at least 12 months. CBD stone recurrence was defined as recurrent stones confirmed by ERCP during the follow-up period. The maximum diameter of the balloon used was 15mm.

CONTACTS AND LOCATIONS:
Overall Officials: Gregorios Gregorios, Director, Study Director — ''Benizelion" General Hospital, Heraklion, Crete
Locations (1):
- ''Benizelion" General Hospital, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: No